CLINICAL TRIAL: NCT00000630
Title: Phase I Safety and Immunogenicity Trial of Vaccinia-HIV Envelope Recombinant Vaccine (HIVAC-1e) in Combination With Soluble Recombinant Envelope Vaccine (gp160; VaxSyn)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Prevention
Other Study IDs: AVEG 002A; 10538 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-27 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Vaccines, Synthetic; Vaccinia Virus; Viral Envelope Proteins; Acquired Immunodeficiency Syndrome; AIDS Vaccines; HIV Seronegativity; HIV Preventive Vaccine
MeSH Terms: conditions — HIV Infections; Vaccinia; Acquired Immunodeficiency Syndrome | interventions — HIVAC-1e; VaxSyn HIV-1 (gp160) vaccine

INTERVENTIONS:
Biological: HIVAC-1e
Biological: gp160 Vaccine (MicroGeneSys)

SUMMARY:
To determine if priming (giving the first vaccination) with a vaccinia recombinant (HIVAC-1e) provides a significant advantage in immunogenicity (production of antibodies) compared to priming with a soluble recombinant protein (gp160); to learn more about the safety of the combination use of the two HIV envelope vaccines utilized in the study.

Recent studies at the AIDS vaccine units have shown the safety of two candidate HIV vaccines, HIVAC-1e and gp160. Specific questions to be addressed in this part of the study include: Does combination vaccination result in a synergistic (added) response not predicted by just the addition of a second vaccination, and does this synergism depend on the unique priming effect of a vaccinia recombinant, or will any combination do?

DETAILED DESCRIPTION:
Recent studies at the AIDS vaccine units have shown the safety of two candidate HIV vaccines, HIVAC-1e and gp160. Specific questions to be addressed in this part of the study include: Does combination vaccination result in a synergistic (added) response not predicted by just the addition of a second vaccination, and does this synergism depend on the unique priming effect of a vaccinia recombinant, or will any combination do?

Volunteers will be randomized to one of four groups. Group A (20 volunteers) will receive gp160 (VaxSyn) followed two months later by a repeat dose. Group B (20 volunteers) will receive VaxSyn followed two months later by HIVAC-1e. Group C (20 volunteers) will receive HIVAC-1e followed two months later by VaxSyn. Group D (10 volunteers) will receive HIVAC-1e followed two months later by HIVAC-1e. For volunteers in Groups A, B, and C who do not react to the initial vaccination, a second attempt to obtain a reaction may be made 7 or more days following the initial inoculation. Per addendum, two additional booster inoculations are given: one at 6 months or later post initial inoculation (Groups A, C, and D receive VaxSyn and Group B receives HIVAC-1e) and another at 12 months or later (all Groups receive VaxSyn).

ELIGIBILITY:
Inclusion Criteria

* Volunteers must be healthy adults without high-risk behavior for HIV-1 infection and with history of smallpox vaccination more than 5 years prior to enrollment.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms and conditions are excluded:

* Identifiable high-risk behavior for HIV infection including active intravenous drug use and multiple sexual partners or sexual contact with high-risk partners within the past 6 months.
* Eczema, active or within the past year.
* Household contact with someone who is pregnant.
* Household contact with children less than 12 years old.
* Household contact with anyone with eczema.
* Household contact with anyone with immunodeficiencies.
* Hypersensitivity to insects.
* Medical or psychiatric conditions that would make compliance unlikely.
* Evidence of depression.

Patients with the following prior conditions are excluded:

* History of immunodeficiency or chronic illness or use of immunosuppressive medications.
* Blood or blood product transfusion within previous six months.
* Eczema, active or within the past year.
* Prior receipt of experimental HIV vaccine. [Specific other requirements are stated elsewhere in the record.]

Prior Treatment:

Excluded within 6 months prior to study entry:

* Blood or blood product transfusions.

Risk Behavior:

Excluded:

* Active intravenous drug use.
* Syphilis, gonorrhea, or any sexually transmitted diseases including chlamydia or pelvic inflammatory disease within the past 6 months.
* More than 2 sexual partners in the past 6 months or sexual contact with a high-risk partner.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35
Dates: Study Completion 1992-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Koff W, Study Chair
Locations (2):
- United States (2):
  - Vanderbilt Univ. Hosp. AVEG, Nashville, Tennessee
  - UW - Seattle AVEG, Seattle, Washington